CLINICAL TRIAL: NCT06919393
Title: "Triple Negative" Adult B-cell Acute Lymphoblastic Leukemia: Molecular Characterization, Identification and New Stratification
Brief Title: "Triple Negative" Adult B-cell Acute Lymphoblastic Leukemia - TRINEG-ALL
Acronym: TRINEG-ALL
Status: Recruiting | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRSTB098
Record Dates: First submitted 2021-02-25; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Leukemia, Lymphoblastic
Keywords: lymphoblastic acute leukemia (LAL); triple negative; B cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh peripheral blood and bone marrow samples will be collected before treatment and/or at relapse.
  Saliva sample will be collected for each enrolled patient. Whenever possible, saliva sample should be collected during treatment, in order to reduce tumor contamination; if not feasible, saliva sample can be collected at patient enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "Triple negative" adul B-cell ALL: Prospective and retrospective cohorts.
  Interventions: Other: "Triple negative" adul B-cell ALL

INTERVENTIONS:
Other: "Triple negative" adul B-cell ALL — Samples will be studied with conventional techniques to classify and define properly the disease: morphology, immunophenotype, immunohistochemistry (IHC), conventional Cytogenetic Fluorescence in Situ Hybridization (FISH) will be used when appropriate.
  ● Isolation of Mononuclear cells
  The following research methodologies will be applied:
  * Next Generation Sequencing
  * Flow cytometry analysis of 3C-up B-ALL top three markers
  * Gene expression profile analysis
  * Copy number Alterations analysis
  * In vitro studies

SUMMARY:
It is a multicenter, non-interventional, non pharmacological, translational, prospective study. Any decision about drug administration is made by the physician based on his clinical judgment in the context of clinical practice, independently from the decision to include the patient in the study.

DETAILED DESCRIPTION:
Survival rates from Acute lymphoblastic leukemia (ALL) have improved dramatically over the past four decades but vary significantly with age. Children treated on modern protocols have survival rates exceeding 90%. Although the remarkable progress made in the treatment of B-Acute lymphoblastic leukemia (B-ALL) in children and, with less efficacy, in adults, several ALL subtypes continue to have a poor prognosis and in a proportion of long-term surviving patients, treatment is responsible for short and long-term toxicities. Consequently, there is a need in improving the molecular dissection of subtypes, identifying genetic alterations that predict the risk of treatment failure and developing novel and targeted therapies. B-ALL patients that doesn't have the most recurrent adult rearrangements (breakpoint cluster region (BCR) - Abelson murine leukemia viral oncogene homolog 1 (ABL1) t(9;22); Transcription Factor 3 (TCF3) - Pre-B-cell leukemia transcription factor 1(PBX1) t(1;19); mixed-lineage leukemia 1 (MLL) - ALL1-fused gene from chromosome 4 (AF4) t(4;11)) are collectively referred to as triple negative (Ph-/-/-) ALL (that represents 61% of adult B-ALL; Roberts KG, J Clinical Oncology 2016). Triple negative ALL is a heterogeneous group of patients; most of these patients have a poor prognosis and miss a target therapy. In the last few years the role of CRLF2 (cytokine receptor-like factor 2; a type I cytokine receptor) gene have become pivotal in ALL, both in adult and paediatric patients. In the last few years the role of CRLF2 (cytokine receptor-like factor 2; a type I cytokine receptor) gene have become pivotal in ALL, both in adult and paediatric patients. CRLF2 is frequently altered in adult B-ALL, especially in Ph-like pts (50-75% of cases) and in Down syndrome ALL (50% to 55%). Alterations that lead, in the majority of cases, to a CRLF2 overexpression. Adult pts with upregulated CRLF2 have poor outcome and novel strategies are needed to improve it.

It is a multicenter, non-interventional, non pharmacological, translational, prospective study. Any decision about drug administration is made by the physician based on his clinical judgment in the context of clinical practice, independently from the decision to include the patient in the study.

The primary objective is the biological characterization of Ph-/-/- ALL, considering CRLF2 overexpression event, in order to define cluster of patients and to assess biomarkers in this subgroup to test new drugs.

The secondary objective is to evaluate if the cytofluorimetric assay - developed on the basis of preliminary data - may be used to detect triple negative subgroups, to provide a rapid, simple and economically viable diagnostic tool to recognize these cases at presentation.

About 60 patients affected by primary or secondary ALL will be enrolled at diagnosis and/or relapse/s.

Patients will be asked to donate part of the Peripheral Blood and Bone Marrow samples, collected according to clinical practice for the management of their disease, for the purposes of this study. A saliva sample will be collected from each patients. Clinical data will be collected in a study dedicated database.

The total duration of the study is 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study;
* Patients with new diagnosis and/or relapse/s of primary or secondary B-ALL;
* Negative for BCR-ABL1 t(9;22); TCF3-PBX1 t(1;19); MLL-AF4 t(4;11) rearrangements;
* Participant is willing and able to give informed consent for participation in the study;
* Male or Female, aged >18 years;
* Availability of clinical data.

Exclusion Criteria:

* Age < 18 years;
* B-ALL positive for BCR-ABL1 t(9;22); TCF3-PBX1 t(1;19); MLL-AF4 t(4;11) rearrangements.

Low blast percentage (<70%) samples could be excluded for molecular evaluations, not for cytofluorimetric analyses;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Ph-/-/- B cell Acute Lymphoblastic Leukemia (see inclusion criteria) will be considered for enrolment. Therefore, patients can be enrolled at diagnosis or relapse/s.
  About 60 patients affected by primary or secondary B-ALL, at diagnosis and/or relapse/s will be enrolled in this study. All suitable prospective fresh PB and/or BM samples will be evaluated with cytofluorimetric panel.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Biological characterization for B-ALL Ph-/-/- subgroup identification | 3 years
  Biological characterization of Ph-/-/- ALL, considering CRLF2 overexpression event, to better define clusters preliminarily identified and to identify biomarkers in these subgroups. Each sample at diagnosis and/or relapse time-point will be sequenced with an RNA-seq capture approach. Through bioinformatic analysis we will identify upregulated CRLF2 samples and associated gene signature. Fusion, mutation identification will integrate expression data.

SECONDARY OUTCOMES:
Correlation, in terms of survival, between identified Ph-/-/- molecular subgroups and eventual novel associated molecular features. | 3 years
  To investigate the association of identified Ph-/-/- molecular subgroups and/or molecular features with the clinical outcome (OS, EFS). To assess if a Ph-/-/- molecular subgroups, identified thanks to our analyses, could be associated with poor prognosis.
Cytofluorimetric evaluation of Ph-/-/- ALL markers as CRLF2, CTGF and CD200. | 3 years
  To evaluate if the cytofluorimetric assay - developed on the basis of preliminary data - may be used to detect triple negative subgroups, to provide a rapid, simple and economically viable diagnostic tool to recognize these cases at presentation. On each enrolled fresh sample cells will be analysed through a B-ALL flow cytometer panel (e.g. CD45, CD19, CD34) to which markers of interest will be added (e.g. CRLF2, CTGF and CD200).
  Their expression in flow cytometry will be compared with the expression obtained from RNA-seq data.
Discover new biomarkers identified Ph-/-/- molecular subgroups | 3 years
  To assess if some molecular feature could be associated to specific Ph-/-/- molecular subgroups. To explore if these biomarkers, detected in some of identified Ph-/-/- molecular subgroups, could be targeted by novel drugs. To evaluate the drug/s effects through sensitivity in vitro/ex vivo tests on B-ALL cell lins and on primary leukemic cells.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, Prof, Study Director — IRST IRCCS
Locations (3):
- Italy (3):
  - Irst Irccs, Meldola, FC
  - Ospedale S. Maria delle Croci RAVENNA, Ravenna, RA
  - Ospedale Infermi, Rimini, RN

IPD SHARING:
Plan to Share IPD: No